CLINICAL TRIAL: NCT06150560
Title: A Phase III, Randomized, Double-Blind, Placebo Controlled Clinical Trial Evaluating the Benefits and Mechanism Of Action Of Angiotensin-II Receptor Blocker On Cardiovascular Remodeling In Patients With Repaired Coarctation Of Aorta
Brief Title: A Study of Angiotensin-II Receptor Blocker on Cardiovascular Remodeling (VALUE Trial)
Acronym: VALUE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-007629; 1R01HL162830-01A1 (NIH)
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Coarctation of Aorta; High Blood Pressure
MeSH Terms: conditions — Aortic Coarctation; Hypertension | interventions — Losartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Losartan Group (Experimental): Subjects with Coarctation of Aorta (COA) and high blood pressure will receive Losartan.
  Interventions: Drug: Losartan
- Amlodipine Group (Active Comparator): Subjects with Coarctation of Aorta (COA) and high blood pressure will receive Amlodipine.
  Interventions: Drug: Amlodipine
- Placebo Group (Placebo Comparator): Subjects with Coarctation of Aorta (COA) and high blood pressure will receive Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — 50mg administered orally once daily for 52 weeks.
  Other Names: Cozaar
  Arms: Losartan Group
Drug: Amlodipine — 5mg Amlodipine administered orally once daily for 52 weeks.
  Arms: Amlodipine Group
Drug: Placebo — Oral capsules that contain no active drug ingredients administered orally once daily for 52 weeks.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness and mechanism of action of Losartan in the treatment of coarctation of aorta.

ELIGIBILITY:
Inclusion Criteria:

* B/S1 hypertension
* SBP 100-139 average based on 3 office measurements.
* Age 18 or Older
* Previous COA Repair

Exclusion Criteria:

* Currently on beta blocker (BB) therapy
* Pregnancy/lactating
* eGFR<30
* Hyperkalemia (serum potassium >5.5mmol/L)
* Severe Aortic or Mitral valve stenosis or regurgitation
* Epicardial CAD diagnosis
* Received antihypertensive medications within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular (LV) Fibrosis | Baseline; Week 52
  LV fibrosis will be measured via indexed Extracellular Volume (iECV) which will be calculated as extracellular volume fraction (ECV%) x LV End Diastolic Volume Index as evaluated during Cardiac Magnetic Resonance Imaging (CMRI).

SECONDARY OUTCOMES:
Change in Exercise Capacity (peak VO2) | Baseline; Week 52
  Change in Exercise Capacity will be evaluated based on peak VO2, measured as milliliters of oxygen per kilogram of body weight per minute (ml/kg/min), during supine bike cardiopulmonary exercise test (Stress Echocardiogram).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, MBBS, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No